CLINICAL TRIAL: NCT01686607
Title: A Multicenter Cohort Study of the Short and Long-term Safety of Micafungin and Other Parenteral Antifungal Agents
Brief Title: Short and Long-term Safety of Micafungin and Other Parenteral Antifungal Agents
Acronym: MYCOS
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Europe B.V. (Industry)
Collaborators: World Health Information Science Consultants, LLC (Other)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: 9463-CL-1401
Record Dates: First submitted 2012-09-13; First posted 2012-09-18 (Estimated); Last update posted 2024-10-21 (Actual); Status verified 2019-05

CONDITIONS: Systemic Fungal Infections
Keywords: Hepatic toxicity; Renal toxicity; Micafungin; Hepatocellular carcinoma; Antifungals (parenteral)
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Caspofungin; Anidulafungin; Fluconazole; Itraconazole; Voriconazole; Amphotericin B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1) parenteral micafungin users: patients who had been treated with parenteral micafungin
  Interventions: Drug: Parenteral micafungin application
- 2) other parenteral antifungal users: patients who had been treated with a parenteral antifungal agent (not micafungin)
  Interventions: Drug: Other parenteral antifungal drugs

INTERVENTIONS:
Drug: Parenteral micafungin application — Parenteral
  Groups: 1) parenteral micafungin users
Drug: Other parenteral antifungal drugs — Parenteral
  Other Names: caspofungin; anidulafungin; fluconazole; itraconazole; voriconazole; amphotericin B (various formulations); 'other antifungals' include the following drugs:
  Groups: 2) other parenteral antifungal users

SUMMARY:
This multicenter observational cohort study proposes to establish the risks of short and long-term outcomes in users of parenteral micafungin and in users of other parenteral antifungal agents from 2005 through 2012 with follow-up until 2017.

DETAILED DESCRIPTION:
All eligible patients treated with a parenteral antifungal agent at any time during the years 2005-2012 in each of the participating hospitals, will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized and treated with parenteral antifungal medication
* first time treatment of the patient with parenteral antifungal in the medical center was anytime from 2005 through 2012

Exclusion Criteria:

* prior diagnosis of hepatocellular carcinoma
* had received parenteral antifungal therapy during the 6 months prior to index hospitalization

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with parenteral antifungals in tertiary referral centers across the United States.
Sampling Method: Non-Probability Sample
Enrollment: 40110 (Actual)
Dates: Start 2012-10-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent hepatic injury or dysfunction | Up to 30 days after termination of the index treatment
  Data will be used of patients treated during the years 2005-2012 with a parenteral antifungal agent in the participating centers.
Treatment-emergent renal failure or dysfunction | Up to 30 days after termination of the index treatment
  Data will be used of patients treated during the years 2005-2012 with a parenteral antifungal agent in the participating centers.
Rehospitalization for the parenteral treatment of fungal infections | Up to 30 days after termination of the index treatment
  Data will be used of patients treated during the years 2005-2012 with a parenteral antifungal agent in the participating centers.
Death from hepatocellular carcinoma (HCC) | Up to 13 years after treatment
  On a long-term basis up to 13 years from 2005-2017.

CONTACTS AND LOCATIONS:
Overall Officials: Lead Investigator, Principal Investigator — WHISCON, LLC
Locations (6):
- United States (6):
  - Site US4, Baltimore, Maryland
  - Site US2, Boston, Massachusetts
  - Site US6, Ann Arbor, Michigan
  - Site US3, Durham, North Carolina
  - Site US5, Philadelphia, Pennsylvania
  - Site US1, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.